CLINICAL TRIAL: NCT05797948
Title: Prospective, Single-center, Single-arm, Open-label Study of Obinutuzumab, Zanubrutinib and Lenalidomide Sequential CD19/CD22 CAR-T in Patients With Relapsed or Refractory B-Cell Non-Hodgkin Lymphoma
Brief Title: GZL Sequential CD19/CD22 CAR-T in Relapsed or Refractory B-cell Non-Hodgkin Lymphoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GZL
Record Dates: First submitted 2023-03-22; First posted 2023-04-04 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-02

CONDITIONS: Relapsed or Refractory B-cell Non-Hodgkin Lymphoma
Keywords: Humanized anti-CD20 monoclonal antibody; BTK Inhibitor; Immunomodulators; CAR-T
MeSH Terms: conditions — Recurrence; Lymphoma, B-Cell | interventions — obinutuzumab; zanubrutinib; Lenalidomide; Azacitidine; Injections; fludarabine; fludarabine phosphate; Cyclophosphamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GZL sequential CD19/CD22 CAR-T (Experimental): Phase I (combined immunotherapy period):
  2-4 cycle of combination chem-free therapy with Obinutuzumab, Zanubrutinib and Lenalidomide . Each cycle is 21 days.
  Phase II (CAR-T therapy):
  CAR-T therapy with AZA + FC (Azacitidine, Fludarabine and Cyclophosphamide) conditioning regimen. Targets of CAR-T cells are CD19/CD22.
  Interventions: Drug: Obinutuzumab; Drug: Zanubrutinib; Drug: Lenalidomide; Drug: CD19/CD22 CAR-T; Drug: Azacitidine For Injection; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Obinutuzumab — Obinutuzumab Injection 1000mg ivgtt C1-C4 d1；
  Other Names: Gazyva
Drug: Zanubrutinib — Zanubrutinib 160mg (2 capsules) oral bid；
  Other Names: Brukinsa
Drug: Lenalidomide — Lenalidomide 25mg (1 capsule) oral C1-C4 d1-d10.
  Other Names: Anxian
Drug: CD19/CD22 CAR-T — Targets of CAR-T cells are tandem CD19/CD22. 1 * 10 ^ 7/kg dual-target CAR-T cells were reinfused with 10%, 30% and 60% of the total dose on d1, d2, d3 respectively.
Drug: Azacitidine For Injection — Azacitidine For Injection 100mg i.h. d1-d5;
  Other Names: Anyve
Drug: Fludarabine — Fludarabine 300mg/m2 ivgtt d3-d5;
  Other Names: Fludara
Drug: Cyclophosphamide — Cyclophosphamide 300mg/m2 ivgtt d3-d5.
  Other Names: Endoxan

SUMMARY:
This study intends to use Obinutuzumab, Zanubrutinib, and Lenalidomide sequential CD19/CD22 CAR-T in the treatment of Relapsed or Refractory B-cell Non-Hodgkin Lymphoma patients. The main purpose of this study is to explore a new treatment mode for R/R B-NHL patients and observe the efficacy and safety of this treatment regimen.

DETAILED DESCRIPTION:
The study will start with 2-4 cycles of combination chem-free therapy with obinutuzumab, zanubrutinib and lenalidomide, followed by sequential CAR-T therapy. CAR-T therapy with AZA + FC (Azacitidine +Fludarabine +Cyclophosphamide) conditioning regimen. Targets of CAR-T cells are CD19/CD22. In this clinical trial, ORR, CRR, OS, PFS, AE and other indicators were used to observe the safety and efficacy of this sequential therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed CD22 + and/or CD19 + aggressive B-cell non-Hodgkin lymphoma (NHL), including the following types as defined by World Health Organization (WHO) 2016:

   Diffuse large B-cell lymphoma (DLBCL); High grade B-cell lymphoma (HGBL); Primary mediastinal large B-cell lymphoma(PMBCL); T cell/histiocyte-rich large B-cell lymphoma (THRBCL); High grade follicular cell lymphoma Grade 3b (3bFL); Mantle cell lymphoma (MCL) except indolent; Other aggressive B-cell lymphomas.
2. Disease refractory to first-line therapy or early relapse within 12 months of last treatment.
3. Relapse or progressive disease (PD) ≥ 3 months after targeted CD19 therapy including CD19 CAR T cells or anti-CD19/anti-CD3.
4. Successful leukapheresis assessment and T-cell preculture.
5. Life expectancy > 3 months.
6. Appropriate organ function:

   Creatinine < 1.6 mg/dL (140 µmol/L) or creatinine clearance ≥ 60ml/min; Alanine aminotransferase (ALT)/aspartate aminotransferase (AST) < 3 × upper limit of normal; Bilirubin < 2.0 mg/dL unless subject has Gilbert 's syndrome (< 3.0 mg/dL); Pulmonary reserve ≤ Grade 1 dyspnea and SPO2 > 91%; Cardiac ejection fraction ≥ 50% in the absence of oxygen, no evidence of pericardial effusion as determined by echocardiogram (ECHO), and no clinically significant electrocardiogram (ECG) findings.
7. Adequate bone marrow reserve was defined as:

   Absolute neutrophil count (ANC) > 1000/mm3; Absolute lymphocyte count (ALC) ≥ 300/mm3; Platelet count ≥ 50,000/mm3. Hemoglobin > 7.0 mg/dL.
8. Measurable or evaluable lesions according to "IWG response criteria for malignant lymphoma" (Cheson 2014).
9. Patients have the ability to understand and are willing to provide written informed consent.

Exclusion Criteria:

1. severe liver and kidney dysfunction (alanine aminotransferase, bilirubin, creatinine > 3 times the upper limit of normal);
2. the presence of structural heart disease, and lead to clinical symptoms or abnormal heart function (NYHA ≥ 2);
3. uncontrolled active infection;
4. the presence of other tumors requiring treatment or intervention;
5. the current or expected need for systemic corticosteroid therapy;
6. pregnant or lactating women.
7. Other psychological conditions that prevent patients from participating in the study or signing informed consent;
8. According to the investigator 's judgment, the subject is unlikely to complete all protocol-required study visits or procedures, including follow-up visits, or fail to meet the requirements for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) after GZL therapy | At the end of GZL therapy (2-4 cycles, each cycle is 21days)
  the rate of patients who achieved CR or PR after GZL therapy
Complete response rate (CRR) after CAR-T | Within 3 months after CAR-T therapy
  the best rate of patients who achieved CR after CAR-T therapy
Progression-free survival (PFS) after CAR-T | up to 24 months after the end of last patient's treatment
  PFS will be assessed from the GZL combination therapy given to date of progression, relapse, death or end of follow-up.

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events, treatment-related adverse events and serious adverse events | Initiation of GZL therapy until 30 days after CAR-T therapy
  The safety and tolerability of the therapeutic regimen measured by the incidence of Treatment-Emergent Adverse Event.
Overall response rate (ORR) after CAR-T | Within 3 months after CAR-T therapy
  The best rate of patients who achieved CR or PR after CAR-T therapy
Overall survival (OS) after CAR-T | up to 24 months after the end of last patient's treatment
  OS will be assessed from the GZL combination therapy given to date of death or end of follow-up.
Duration of Response(DOR) after CAR-T | up to 24 months after the end of last patient's treatment
  DOR will be assessed from the date of CAR-T infusion to the date of progression, relapse, death or end of follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
All the data would be available at the First Affiliated Hospital and other researchers after the end of the study.
Supporting Information: Study Protocol, SAP
Time Frame: after the end of the study